CLINICAL TRIAL: NCT03799731
Title: Open, Non Controlled, Parallel Cohorts, Multicenter, Phase 2A Study for Evaluation of the Antitumor Activity of GM102 Single Agent and in Combination With Chemotherapy in Patients With Locally Advanced Or Metastatic Colorectal Cancer
Brief Title: Study for Evaluation of Murlentamab (GM102) Anti-tumoral Activity in Colorectal Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GamaMabs Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C201
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort I: GM102 single agent (Experimental): GM102 will be intravenously administered at the dose of 7 mg/kg on Days 1, 8, 15 and 22 of each 28-day cycle
  Interventions: Drug: GM102
- Cohort II: GM102 + trifluridine/tipiracil (Experimental): GM102 will be intravenously administered at the dose of 7 mg/kg on Days 1, 8, 15 and 22, and trifluridine/tipiracil will be orally administered at the dose of 35 mg/m² twice daily on Days 1 to 5 and days 8 to 12 of each 28-day cycle
  Interventions: Drug: GM102; Drug: Trifluridine/Tipiracil
- Cohort II expansion: GM102 + trifluridine/tipiracil (Experimental): GM102 will be intravenously administered at the dose of 7 mg/kg on Days 1, 8, 15 and 22, after a loading dose of 10 mg/kg q1w during 28-day cycle 1, and trifluridine/tipiracil will be orally administered at the dose of 35 mg/m² twice daily on Days 1 to 5 and days 8 to 12 of each 28-day cycle
  Interventions: Drug: Trifluridine/Tipiracil; Drug: GM102 expansion

INTERVENTIONS:
Drug: GM102 — GM102 7 mg/kg weekly
  Arms: Cohort I: GM102 single agent; Cohort II: GM102 + trifluridine/tipiracil
Drug: Trifluridine/Tipiracil — Lonsurf 35 mg/m² twice daily during 10 days per cycle
  Other Names: Lonsurf
  Arms: Cohort II expansion: GM102 + trifluridine/tipiracil; Cohort II: GM102 + trifluridine/tipiracil
Drug: GM102 expansion — GM102 7 mg/kg weekly after a loading dose of 10 mg/kg q1w during 28-day cycle 1
  Arms: Cohort II expansion: GM102 + trifluridine/tipiracil

SUMMARY:
Phase 2A study, assessing the antitumor activity and the safety profile of GM102, a new compound (monoclonal antibody), administered alone or in combination with chemotherapy in patients with locally advanced or metastatic colorectal cancer. The primary objective of the study is to evaluate the antitumor activity of GM102 single agent and in combination with trifluridine/tipiracil.

DETAILED DESCRIPTION:
GM102 is a humanized low fucose monoclonal antibody with a high affinity to AMHRII receptor (fetal receptor mediating the activity of AMH, reexpressed in a variety of solid tumors). GM102 acts through engagement of immune cells (macrophages, natural killer (NK) cells) to trigger ADCC (antibody dependent cellular cytotoxicity) and phagocytosis of tumor cells.

AMRHII expression was found in 73% of primary colorectal tumors tested.

Advanced/metastatic colorectal cancer (CRC) remains an unmet need disease, with few therapeutic options beyond two or three lines of therapy.

CRC is characterized by a tumor microenvironment (TME) particularly rich in macrophages and more specifically macrophages capable of tumor phagocytosis. The pattern of the TME remains a major prognostic factor in the metastatic setting.

C201 consists in two parallel cohorts and an expansion of cohort II for patients with advanced or metastatic colorectal cancer in two different settings of the disease:

* Cohort I (GM102 as a single agent) in refractory patients, having exhausted all therapeutic options. Patients will receive GM102 alone at the dose of 7 mg/kg administered by intravenous infusion at Day 1, Day 8, Day 15 and Day 22 of each 28-day cycle
* Cohort II (GM102 in combination with trifluridine/tipiracil) in patients candidate to receive single agent trifluridine/tipiracil, after at least two lines of treatment for the advanced or metastatic disease. Patients will receive GM102 at the dose of 7 mg/kg administered by intravenous infusion at Day 1, Day 8, Day 15 and Day 22 and trifluridine/tipiracil at 35 mg/m² per dose twice daily orally administered on Days 1 to 5 and Days 8 to 12 of each 28-day cycle.
* Cohort II expansion (GM102 in combination with trifluridine/tipiracil) same as cohort II except a loading dose of 10 mg/kg q1w during 28-day cycle 1

Patients will be treated with GM102 (Cohort I) or GM102 and trifluridine/tipiracil (Cohort II and Cohort II expansion) until confirmed progression or toxicity.

A Trial Steering Committee (TSC) will analyze and qualify GM102 activity and toxicities and will provide recommendations on the Investigational Medicinal Product (IMP) continuation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or locally advanced colorectal adenocarcinoma.
* Having failed the previous line of treatment for locally advanced or metastatic disease and having received at least two systemic chemotherapy regimens for metastatic colorectal cancer; adjuvant regimen can be considered as one chemotherapy regimen for metastatic disease if the participant had disease recurrence within 6 months of completion.
* At least one of the tumor sites amenable to core needle biopsy (may not be the site of disease for measuring antitumor response). Patient must agree to this pre-treatment biopsy and on the principle of a second biopsy under treatment; however, if eventually the second biopsy cannot be performed, patients will continue on the study and will be considered evaluable for efficacy.
* Available archived CRC tumor tissue sample
* At least one measurable lesion (superior or equal to 1.0 cm longest diameter or superior or equal to 1.5 cm in short axis for malignant lymph nodes) based on RECIST (Response Evaluation Criteria in Solid Tumors) 1.1 on the screening CT-scan.
* Written Informed Consent forms signed.
* Willing and able to comply with the trial requirements.
* Covered by healthcare insurance in accordance with local requirements.
* For cohort I (single agent GM102) only: refractory patients, having exhausted all therapeutic options.
* For cohort II (GM102 in combination with trifluridine/tipiracil) only: patients eligible for trifluridine/tipiracil who have been previously treated with, or are not considered candidates for, available therapies including fluoropyrimidine-, oxaliplatin- and irinotecan-based chemotherapies, anti-Vascular Endothelial Growth Factor (anti-VEGF) agents, regorafenib and anti-Epithelial Growth Factor Receptor (anti-EGFR) agents. Patients must have received at least 2 prior lines of standard chemotherapy for metastatic CRC.

Exclusion Criteria:

* Age < 18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status superior or equal to 2.
* Life expectancy < 12 weeks.
* Major surgery or radiotherapy within 21 days prior to Cycle 1 Day 1 or anticipation of needing such procedure while receiving study treatment.
* Known or symptomatic brain metastasis (other than totally resected or previously irradiated and non-progressive/relapsing) or lepto-meningeal carcinomatosis.
* Concurrent treatment with any other anticancer therapy (or investigational agent) or received any anticancer therapy (or investigational agent) within 4 weeks prior to first treatment.
* Known severe anaphylactic or other hypersensitivity reactions to Investigational Medicinal Product (IMP) and/or its excipients.
* Unresolved toxicity superior or equal to Grade 2 according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 attributed to any prior therapies (excluding anemia, alopecia, skin pigmentation, and platinum induced neurotoxicity).
* Serious concomitant illness, e.g. active infection requiring systemic antibiotic, antifungal or antiviral drug, or physical examination or laboratory abnormalities, that, in the opinion of the Investigator, would compromise protocol objectives.
* Poor bone marrow reserve as defined by white blood cell < 3.0 x 10E9/L, neutrophils < 1.5 x 10E9/L or haemoglobin < 9.0 g/dL or platelet count < 100 x 10E9/L.
* Poor organ function as defined by any one of the following: serum creatinine > 1.5 x upper limit of normal (ULN), total bilirubin > 1.5 x ULN or > 2.5 x ULN if due to Gilbert's syndrome, AST and ALT > 2.5 x ULN in the absence of liver metastasis or > 5 x ULN in case of documented liver metastasis.
* Severe New York Heart Association (NYHA) III and IV heart failure.
* Pregnancy or breastfeeding.
* Patient with reproductive potential who does not agree to use an accepted highly effective method of contraception - per investigator's judgment - during the study period and for at least 6 months following completion of study treatment.
* Patient deprived of liberty by a judicial or administrative decision, patient admitted to a social institution or who is under a measure of legal protection, patient hospitalized without consent or who is in an emergency situation.
* Known allergy to rodents.
* Patients positive to Covid-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Through study completion, an average 1 year
  ORR from the end of cycle 2 and subsequently confirmed at least 4 weeks later using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
Progression Free Survival (PFS) at 6 months | 6 months after the first infusion
  Proportion of patients without documented progression at 6 months

SECONDARY OUTCOMES:
Immune Overall Response Rate (iORR) | Through study completion, an average 1 year
  ORR using immune Response Evaluation Criteria In Solid Tumors (iRECIST)
Clinical Benefit Rate (CBR) | up to 4 months
  CBR at 8 and 16 weeks defined as the number of non-progressors using RECIST 1.1 and iRECIST criteria
Tumor Growth Rate (TGR) before and under treatment | up to 2 months
  Percentage of variation in TGR
Progression Free Survival (PFS) | Through study completion, an average 1 year
  Time elapsed from the date of first infusion to the date of documented progression or death
Overall Survival (OS) | Through study completion, an average 1 year
  Time elapsed from the date of first infusion to the date of death
Incidence of Serious Adverse Event (SAE) and Treatment Emergent Adverse Event (TEAE) | Through study completion, an average 1 year
  Number of events
Pharmacodynamics evaluation | Up to 2 months
  Tumor Immune MicroEnvironment analysis and evolution changes: quantity/density and quality of immune cells
Exposure to murlentamab | At days 1 and 15 of cycles 1, 2 (each cycle is 28 days) and End of Treatment for cohort I and II, an average of one year; days 1, 8,15 and 22 of cycles 1, 2 (each cycle is 28 days) and End of Treatment for cohort II expansion, an average of one year
  PK parameters analysis
Exposure to trifluridine | At days 1 and 15 of cycles 1, 2 (each cycle is 28 days) and End of Treatment, an average of one year
  Trifluridine plasma concentrations only for cohort II
Evidence of anti-murlentamab antibodies (ADA) | Baseline, beginning of every even cycle in pre-dose (each cycle is 28 days) and at the End of Treatment, an average of one year
  Presence of ADA
AMHRII (Anti-Mullerian Hormone type II receptor) expression | Up to 2 months
  AMHRII membrane expression in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Eric Van Cutsem, MD, Principal Investigator — UZ Leuven, Belgium
Locations (5):
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Gasthuisberg, Ghent
  - UZ Leuven, Leuven
- Czechia (2):
  - University Hopistal Olomouc, Olomouc
  - University Hospital Motol, Prague

IPD SHARING:
Plan to Share IPD: No